



## THE ASSESSMENT OF CEREBRAL HAEMODYNAMICS IN PATIENTS WITH TRANSIENT ISCHAEMIC ATTACK: A TRANSCRANIAL DOPPLER STUDY

## **CONSENT FORM (VOLUNTEER)**

| Participant Study ID Number: | | Please initial |
|---|---|---|
| 1. | I confirm that I have read and understand the Information Leaflet ( <i>Version xx, Dated xx/xx/xxxx</i> ) for the above study, and have had the opportunity to ask questions and have had these answered satisfactorily. | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving reason, without my medical care or legal rights being affected. | |
| 3. | I agree that if I decide to withdraw prior to the completion of the study, any health information and data that has been collected up until my point of withdrawal will be retained for the final analysis. | |
| 4. | I understand that my GP will be informed about my participation in this study, and by signing this consent form I am granting permission for this. | |
| 5. | I understand that if there are any incidental findings as a result of participation in this study, my GP will be informed to investigate this further and by signing this consent form I am granting permission for this. | |
| 6. | I understand that data collected during the study may be looked at by responsible individuals from the study team, the sponsor (University of Leicester), NHS Trust or from regulatory authorities, where it is relevant to taking part in this research. I give permission for these individuals to have access to my records. | |
| 7. | I understand that my personal data will be treated with confidentiality and stored as described in the Information Leaflet ( <i>Version xx, Dated xx/xx/xxxx</i> ). | |
| 8. | I understand that my anonymised research data may be shared with researchers from other departments or Universities undertaking similar research, and I grant my permission for this. | |
| 9. | I would like a lay summary of the results of the study sent to me by post or email | □ N □ |
| | at the end of the study (Please tick) Post [ | ☐ Email ☐ |
| 10. | I agree to take part in the above study. | |
| Par | ticipant Name: Signature: | |
| Res | earcher Name: Date: Signature:<br>e: 1 for participant, 1 (original) to be retained in the trial master file) | |